CLINICAL TRIAL: NCT02359357
Title: A Phase 1, Randomised, Double-Blind, Placebo-Controlled, Dose-Escalation First-Time-in-Human Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of Single and Repeat Oral Doses of FDL169 in Healthy Volunteers
Brief Title: FTIH - Single and Repeat Oral Doses of FDL169 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: FDL169-2014-01; RD 674/25728 (Other: Sponsor)
Record Dates: First submitted 2015-01-13; First posted 2015-02-10 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (22):
- Placebo single dose (Placebo Comparator): Placebo administered as a single dose
  Interventions: Drug: Placebo
- Single dose (Dose level 1) (Experimental): FDL169 (Dose level 1) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 2) (Experimental): FDL169 (Dose level 2) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 3) (Experimental): FDL169 (Dose level 3) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 4) (Experimental): FDL169 (Dose level 4) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 5) (Experimental): FDL169 (Dose level 5) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 6) (Experimental): FDL169 (Dose level 6) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 7) (Experimental): FDL169 (Dose level 7) administered as a single dose
  Interventions: Drug: FDL169
- Single dose (Dose level 8) (Experimental): FDL169 (Dose level 8) administered as a single dose
  Interventions: Drug: FDL169
- Additional single dose 1 (Experimental): Single dose of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Additional single dose 2 (Experimental): Single dose of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Additional single dose 3 (Experimental): Single dose of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Additional single dose 4 (Experimental): Single dose of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Food effect - fasted (Experimental): Single dose of FDL169 in fasted conditions
  Interventions: Drug: FDL169
- Food effect - fed (Experimental): Single dose of FDL169 in fed conditions
  Interventions: Drug: FDL169
- Placebo - multiple dose (Placebo Comparator): Repeat doses of placebo
  Interventions: Drug: Placebo
- Multiple dose - Dose level 1 (Experimental): Repeat doses of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Multiple dose - Dose level 2 (Experimental): Repeat doses of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Multiple dose - Dose level 3 (Experimental): Repeat doses of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Multiple dose - Dose level 4 (Experimental): Repeat doses of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Multiple dose - additional dose level 1 (Experimental): Repeat doses of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169
- Multiple dose - additional dose level 2 (Experimental): Repeat doses of FDL169 to be administered at a dose level to be determined (up to Dose level 8)
  Interventions: Drug: FDL169

INTERVENTIONS:
Drug: FDL169
  Arms: Additional single dose 1; Additional single dose 2; Additional single dose 3; Additional single dose 4; Food effect - fasted; Food effect - fed; Multiple dose - Dose level 1; Multiple dose - Dose level 2; Multiple dose - Dose level 3; Multiple dose - Dose level 4; Multiple dose - additional dose level 1; Multiple dose - additional dose level 2; Single dose (Dose level 1); Single dose (Dose level 2); Single dose (Dose level 3); Single dose (Dose level 4); Single dose (Dose level 5); Single dose (Dose level 6); Single dose (Dose level 7); Single dose (Dose level 8)
Drug: Placebo
  Arms: Placebo - multiple dose; Placebo single dose

SUMMARY:
To determine the safety and tolerability of single and multiple escalating doses of FDL169 in healthy male subjects.

DETAILED DESCRIPTION:
This study is the first time in human study and consists of two parts.

Part 1A:

Part 1 of the study is a randomised, double-blind, placebo-controlled, dose-escalation, first-time-in-human study to assess the safety, tolerability and PK profiles following single oral administrations of FDL169 to healthy male volunteers. Sixty-four (64) male subjects (8 per cohort) will be included in Part 1 of the study. Up to eight dose levels of FDL169 are planned to be tested in Part 1 of the study.

Part 1B:

Open label. Following completion of Part 1A of the study, an additional cohort of 8 subjects will receive a single dose of FDL169 in both fasted and fed states

Part 2:

Part 2 of the study is a randomised, double-blind, placebo-controlled, dose-escalation study to assess the safety, tolerability and PK profiles following multiple oral administrations of FDL169 to healthy male subjects. Forty-eight male subjects, in cohorts of twelve, will be included in Part 2 of the study. It is planned to test up to four dose levels of FDL169 in Part 2.

ELIGIBILITY:
Inclusion Criteria:

Healthy male subjects aged 18 to 45 years who fulfil standard safety screening assessments for the study (haematology/biochemistry, urinalysis, 12-lead electrocardiogram (ECG), vital signs and oral temperature) and who in the opinion of the Investigator, are medically suitable to participate in the study. Male subjects and their partners must be willing to use an effective method of contraception from first dose of investigational medicinal product (IMP) and for 3 months after the last dose of IMP.

Exclusion Criteria:

1. Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months.
2. Subjects who have history or presence of clinically significant cardiovascular, pulmonary, renal, hepatic, haematologic, gastrointestinal (endocrine or immunologic disease), at Screening.
3. Donation of 500 mL or more blood within the previous 3 months.
4. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 21 days (or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Flatley Discovery Labs Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
5. Smoking or use tobacco products or substitutes equivalent to > 15 cigarettes/day.
6. Any subject attempting to father a child within 3 months of their Follow-Up Visit.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Part 1A: safety and tolerability for 48 h following single oral doses of FDL169 (Vital signs, electrocardiogram (ECG), safety laboratory data and adverse events (AEs) | Multiple points from screening to follow-up (up to 28 days)
  Vital signs, electrocardiogram (ECG), safety laboratory data and adverse events (AEs)
Part 1B: food effect on the tolerability of FDL169 for 48 h following a single dose | Multiple points from screening to follow-up (up to 42 days)
  Vital signs, ECG, safety laboratory data and AEs
Part 2: safety and tolerability following multiple oral doses of FDL169 (assessed throughout dosing and for 24 h post-final dose) (Vital signs, ECG, safety laboratory data and AEs) | Multiple points from screening to follow-up (up to 42 days)
  Vital signs, ECG, safety laboratory data and AEs
Part 1B: food effect on the pharmacokinetics of FDL169 for 48 h following a single dose | Multiple points from pre-dose to 48 h post-dose
  Pharmacokinetic parameters: Cmax, tmax, lambdaz, t1/2, AUC(0-t), AUC(0-tau), AUC (0-inf) CL/F and AUC%extrapolated

SECONDARY OUTCOMES:
Part 1: pharmacokinetic profile for 48 h following single oral doses of FDL169 | Multiple points from pre-dose to 48 h post-dose
  Pharmacokinetic parameters: Cmax, tmax, lambdaz, t1/2, AUC(0-t), AUC(0-tau), AUC (0-inf) CL/F and AUC%extrapolated
Part 2: pharmacokinetic profile following multiple oral doses of FDL169 (assessed throughout dosing and for 24 h post-final dose) | Multiple points from pre-dose to 24 h post-dosing on Day 14
  Pharmacokinetic parameters: Cmax, tmax, lambdaz, t1/2, AUC(0-t), AUC(0-tau), AUC (0-inf) CL/F and AUC%extrapolated

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, MD, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, Wales, United Kingdom